CLINICAL TRIAL: NCT00012935
Title: Treatment Decision Intervention for Veterans With Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: PCI 99-159
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Insemination, Artificial, Heterologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: Help with decision making on prostate cancer treatment

INTERVENTIONS:
Behavioral: Help with decision making on prostate cancer treatment

SUMMARY:
Newly diagnosed localized prostate cancer patients face difficult decisions about treatment and management; including radiation therapy, radical prostatectomy, brachytherapy, and observation. Previous studies have cited patient preference and physician recommendation for treatment as major roles in treatment decisions.

DETAILED DESCRIPTION:
Background:

Newly diagnosed localized prostate cancer patients face difficult decisions about treatment and management; including radiation therapy, radical prostatectomy, brachytherapy, and observation. Previous studies have cited patient preference and physician recommendation for treatment as major roles in treatment decisions.

Objectives:

This grant will be used to develop and evaluate a decision analysis based intervention to improve decision-making among veterans with newly diagnosed localized prostate cancer. While the ultimate goal of this study is to improve decision-making among these patients, factors influencing physician recommendations for treatment will be sought. The former will be achieved by evaluating the efficacy of providing physicians with information incorporating patient preference for alternative health states with probabilities of treatment outcomes. Factors influencing physician recommendations for treatment will be determined through qualitative interviews with physicians.

Methods:

Patients were accrued at the VA Chicago Health Care System Lakeside Urology Clinic. Upon consent for participation in the study, comorbidities, histologic grade of the biopsy, and age were obtained for 13 patients with newly diagnosed localized prostate cancer. Using a standard gamble technique, interviewers obtained patient utilities for 5 distinct health states related to prostate cancer treatment. Clinical and pathologic characteristics were incorporated into the decision analytic model, and the derived quality-adjusted life expectancies (QALEs) were shared with the treating urologist before patient-physician discussion of treatment options. The feasibility of the decision analytic intervention and unbiased estimates of the impact of the intervention was evaluated. The long-range objective of this proposal is to design an intervention for veterans that increases physician understanding of patient treatment preferences and patient understanding of choices in prostate cancer treatment.

Status:

Completed

ELIGIBILITY:
Inclusion Criteria:

1) biopsy confirmed diagnosis of localized prostate cancer; 2) newly diagnosed-no prior treatment (including watchful waiting) or discussion with their prior physicians about treatment options; 3) no previous neoplasms in the last five years, with the exception of basal cell cancer of the skin; 4) speak english; 5) no major psychiatric disorder that would preclude their participation; 6) be between 50 and 80 years of age.

Exclusion Criteria:

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Study Completion 2001-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles L. Bennett, MD PhD MPP, Principal Investigator — Jesse Brown VA Medical Center Community-Based Outpatient Clinic Lake Side Divison, Chicago, IL; Sara J. Knight, PhD, Principal Investigator — Jesse Brown VA Medical Center Community-Based Outpatient Clinic Lake Side Divison, Chicago, IL
Locations (1):
- Jesse Brown VA Medical Center Community-Based Outpatient Clinic Lake Side Divison, Chicago, IL, Chicago, Illinois, United States

REFERENCES:
- [Result] Knight SJ, Nathan DP, Siston AK, Kattan MW, Elstein AS, Collela KM, Wolf MS, Slimack NS, Bennett CL, Golub RM. Pilot study of a utilities-based treatment decision intervention for prostate cancer patients. Clin Prostate Cancer. 2002 Sep;1(2):105-14. doi: 10.3816/cgc.2002.n.012. PMID 15046701